CLINICAL TRIAL: NCT01555112
Title: A Phase I/II, Open Labeled, Uncontrolled, Single Center Study of Topical AS101 for External Genital Warts
Brief Title: Safety and Efficacy Study to Test Topical AS101 for External Genital Warts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMAS Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS101-IL#001
Record Dates: First submitted 2012-03-11; First posted 2012-03-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Wart; External Genital Organs; Condyloma Acuminata
MeSH Terms: conditions — Warts | interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical AS101 (Experimental): 15% AS101 ointment applied twice a day for treatment of external genital warts.
  Interventions: Drug: Topical AS101

INTERVENTIONS:
Drug: Topical AS101 — AS101 15% ointment will be applied topically twice daily on external genital warts for up to 16 weeks.

SUMMARY:
The purpose of this study is to determine whether the improved topical ointment formulation, AS101, is safe and effective in the treatment of external genital warts in females.

DETAILED DESCRIPTION:
Human papillomavirus (HPV)-induced condyloma acuminata (CA), commonly known as anogenital or genital warts, is among the most common sexually transmitted diseases. There are a wide variety of available treatments of genital warts, but none are considered completely effective. It has been suggested that AS101 works by stimulating the innate and acquired arms of the immune system.

In previous proof-of-concept clinical study AS101 topical cream was tested on HPV warts and shown cure in high percentages. However the cream formulation was unstable therefore a new formulation was developed mainly for the carrier. In this study the improved AS101 ointment will be tested in female patients with external genital warts in an open study to assess its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age and in good health;
* Must sign an ethics committee approved informed consent form and be able to adhere to study visits and protocol requirements;
* Women must agree to avoid sexual contact while the ointment is on their skin;
* All study participants who are sexually active must use a barrier protection method of contraception such as condom in addition to another birth control measure such as oral contraceptives, intrauterine device, spermicide or surgical sterilization during treatment and for 60 days after completion of treatment;
* Patients with first clinical diagnosis of external genital warts, in the external genitalia including vulva (labia minora and majora), inguinal folds, pubic area, perineum, perianal, or buttocks areas;
* A minimum of one lesion and a maximum of 10 lesions identified at study entry, and the maximum diameter of the largest wart is no larger than 10 mm;
* Papanicolaou smears must be obtained in all females within 12 months of Day 1 and be negative for evidence of high grade intraepithelial neoplasia. Women with high grade intraepithelial neoplasia on cytology will be eligible if subsequent colposcopy with biopsy of suspicious area is negative for high grade squamous intraepithelial lesions (Grade 2 or 3). Atypia, HPV effect, and low grade intraepithelial lesions (Grade 1) are acceptable.

Exclusion Criteria:

* Participation in an investigational trial within 30 days prior to Day 1;
* Use of systemic steroids within 30 days of Day 1;
* Previous participation in a trial investigating AS101 for any indication.
* Any prior treatment for genital warts prior to participation;
* Topical and systemic immunosuppressive or immunomodulatory medications (including corticosteroids) within 30 days prior Day 1, and while on study;
* Known history of HIV, HBV and HCV viral infection.
* Current active infection with herpes genitalis or history of herpes genitalis infection within the last 30 days prior to Day 1 (patients on long-term suppressive antiviral therapy are eligible);
* Current and/or recurrent pathologically relevant genital infections other than genital warts;
* Diagnosis of high-grade cervical dysplasia;
* Internal anogenital, vaginal, urethral and cervical warts requiring treatment;
* Chronic or acute skin condition that might interfere with the evaluation of the treatment or study drug effect;
* Cutaneous surgery, including cryosurgery, to genital area within 30 days of Day 1;
* Screening laboratory tests results from a complete blood count (CBC), chemistry panel, urine pregnancy test and urinalysis obtained during screening (Day -14 to Day 0):

  * Must be within the site laboratory's defined normal reference ranges, and/or according to the Investigator's decision;
  * Urine pregnancy test in females of childbearing potential must be negative;
  * Inadequate renal function: Serum Creatinine > 2.0mg/dL (> 2.0 ULN);
  * Inadequate liver function: Serum (total) Bilirubin > 2 mg/dl or ALT and/or AST greater than two times the upper limit of the reference range.
* Uncontrolled infection or acute severe febrile illness;
* Diagnosed as having uncontrolled autoimmune disease;
* Pregnant or lactating;
* Current drug or alcohol abuse that may interfere with the objectives of the study;
* Known allergy to AS101 or any component of the investigational formulation;
* Subjects with any other clinically significant medical condition, psychiatric condition or laboratory abnormality which would, in the judgment of the Investigator, interfere with the subject's ability to participate in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The number of patients with Adverse Events and their severity | up to 16 weeks

SECONDARY OUTCOMES:
Number of patients with complete and partial clearance of external genital warts | 16 weeks
Number of warts that were completely or partially cleared | 16 weeks
Time to complete clearance | 16 weeks
Recurrence rate in treatment area | 3 months follow up
Time to recurrence | 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Shabtai Romano, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Gynecology department, Haemek MC, Afula, Israel